CLINICAL TRIAL: NCT03295058
Title: Outcome of Peripheral Blood Allogenic Stem Cell Transplantation Using Non-anti Thymocyte Globulin (ATG ) Conditioning Regimens in Severe Aplastic Anemia Patients
Brief Title: Peripheral Blood Allogenic Stem Cell Transplantation Using Non-anti Thymocyte Globulin Regimens in Severe Aplastic Anemia Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nourhan Taleb Mohamed, Principal Investigator, Assiut University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPALLSCT
Record Dates: First submitted 2017-09-24; First posted 2017-09-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Severe Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Intervention Model Description: severe aplastic anemia patients will receive two different conditioning regimens before doing allogenic stem cell transplantation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non ATG regimen (Experimental): the first 50% of patients will receive Fludarabine + cyclophosphamide prior to hematopoietic cell transplantation. GVHD Prophylaxis: Cyclosporine A All the patient will do allogenic stem cell transplantation from peripheral blood
  Interventions: Drug: Non ATG Conditioning regimen; Drug: GVHD Prophylaxis; Procedure: Allogenic Stem Cell Transplantation
- ATG regimen (Experimental): the other 50% will receive Cyclophosphamide + ATG prior to hematopoietic cell transplantation. GVHD Prophylaxis: Cyclosporine A All the patient will do allogenic stem cell transplantation from peripheral blood
  Interventions: Drug: GVHD Prophylaxis; Procedure: Allogenic Stem Cell Transplantation; Drug: ATG conditioning regimen

INTERVENTIONS:
Drug: Non ATG Conditioning regimen — 50% of the patients will receive Fludarabine + cyclophosphamide (F-araA 120 mg/m2 total dose for 3 days (d-3,-2,-1) over 1 h infusion and cyclophosphamide 25 mg/kg/d (d-5 to d-2) for 4 days over 1-h infusion prior to hematopoietic cell transplantation , then post transplant cyclophosphamide dose 50 mg/kg on days +3 and +4
  Arms: Non ATG regimen
Drug: GVHD Prophylaxis — Cyclosporine A (CsA 3 mg/kg) start day +5
Procedure: Allogenic Stem Cell Transplantation — using peripheral blood stem cells
Drug: ATG conditioning regimen — the other 50% of the patients will receive Cyclophosphamide + ATG
  Arms: ATG regimen

SUMMARY:
Aplastic anemia is a syndrome of bone marrow failure characterized by peripheral pancytopenia and marrow hypoplasia.The theoretical basis for marrow failure includes primary defects in or damage to the stem cell or the marrow microenvironment

DETAILED DESCRIPTION:
The distinction between acquired and inherited disease may present a clinical challenge, but more than 80% of cases are acquired.

Therapy for aplastic anemia may consist of supportive care only, immunosuppressive therapy, or hematopoietic cell transplantation. Severe and very severe aplastic anemia have a high mortality rate with supportive care alone .

The British Committee for Standards in Haematology recommends treating infection or uncontrolled bleeding before administering immunosuppressive therapy, including in patients scheduled for hematopoietic cell transplantation. The Pediatric Haemato-Oncology Italian Association recommends hematopoietic cell transplantation from a matched sibling donor for severe aplastic anemia, and if a matched donor is not available, options include immunosuppressive therapy or unrelated donor hematopoietic cell transplantation.

Human leukocyte antigen (HLA)-matched sibling-donor hematopoietic cell transplantation is the treatment of choice for a young patient with severe or very severe aplastic anemia , being generally accepted for patients younger than 40 years.

Recent years have seen increasing the use of hematopoietic cells other than bone marrow (BM). These alternative graft sources include peripheral blood progenitor cells and granulocyte colony stimulating factor (G-CSF) bone marrow (G-BM). Several groups have demonstrated that peripheral blood progenitor cell transplantation has faster neutrophil and platelet engraftment compared to BM in patients with hematologic malignancies ; however, most adult studies also report an increase in chronic GVHD (cGVHD) Some adult studies describe improved survival with peripheral blood progenitor cells in adult recipients although survival generally was no different in those with standard-risk disease .

Cyclophosphamide (Cy)/anti-thymocyte globulin (ATG) is considered the standard conditioning regimen for patients with severe aplastic anemia undergoing hematopoietic cell transplantation from a HLA matched sibling donor, The introduction of a fludarabine (F-araA) based reduced intensity conditioning regimen has extended the availability of hematopoietic cell transplantation to patients who are older, heavily transfused and having delayed treatment from the time of diagnosis with HLA matched related/unrelated donors.

The addition of F-araA to the conditioning regimen has been shown to provide additional immunosuppression for engraftment without increasing toxicity in patients undergoing hematopoietic cell transplantation .

Also, conditioning with F-araA and Cy is associated with improved long-term survival compared to a historical cohort receiving Cy/ATG regimen in patients with severe aplastic anemia undergoing hematopoietic cell transplantation .

Adequate post transplantation immunosuppression is important not only for the prevention of GVHD, but also to secure adequate suppression of the host immune system and prevention of graft rejection. The administration of CsA alone or with or without short-course methotrexate or steroid should be considered the standard post transplantation immunosuppression. In addition to possibility of use of other immunosuppressive agents, including the use of mycophenolate mofetil, particularly in patients with renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* All patients with severe and very severe aplastic anemia for stem cell therapy.

Exclusion Criteria:

1- Contraindication to stem cell transplantation. 2 - Patients associated co-morbidities.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Overall Survival rate | two years

SECONDARY OUTCOMES:
GVHD occurrence (Acute or Chronic), engraftment and transplant related mortality | two years
Relapse rate | two years
Progression free survival | two years

REFERENCES:
- [Background] Killick SB, Bown N, Cavenagh J, Dokal I, Foukaneli T, Hill A, Hillmen P, Ireland R, Kulasekararaj A, Mufti G, Snowden JA, Samarasinghe S, Wood A, Marsh JC; British Society for Standards in Haematology. Guidelines for the diagnosis and management of adult aplastic anaemia. Br J Haematol. 2016 Jan;172(2):187-207. doi: 10.1111/bjh.13853. Epub 2015 Nov 16. No abstract available. PMID 26568159
- [Background] George B, Mathews V, Viswabandya A, Abraham A, Ganapule A, Fouzia NA, Korula A, Lakshmi KN, Chandy M, Srivastava A. Immunosuppressive Therapy and Bone Marrow Transplantation for Aplastic Anaemia--The CMC Experience. J Assoc Physicians India. 2015 Mar;63(3 Suppl):36-40. PMID 26529866
- [Background] Barone A, Lucarelli A, Onofrillo D, Verzegnassi F, Bonanomi S, Cesaro S, Fioredda F, Iori AP, Ladogana S, Locasciulli A, Longoni D, Lanciotti M, Macaluso A, Mandaglio R, Marra N, Martire B, Maruzzi M, Menna G, Notarangelo LD, Palazzi G, Pillon M, Ramenghi U, Russo G, Svahn J, Timeus F, Tucci F, Cugno C, Zecca M, Farruggia P, Dufour C, Saracco P; Marrow Failure Study Group of the Pediatric Haemato-Oncology Italian Association. Diagnosis and management of acquired aplastic anemia in childhood. Guidelines from the Marrow Failure Study Group of the Pediatric Haemato-Oncology Italian Association (AIEOP). Blood Cells Mol Dis. 2015 Jun;55(1):40-7. doi: 10.1016/j.bcmd.2015.03.007. Epub 2015 Mar 31. PMID 25976466
- [Background] Socie G. Allogeneic BM transplantation for the treatment of aplastic anemia: current results and expanding donor possibilities. Hematology Am Soc Hematol Educ Program. 2013;2013:82-6. doi: 10.1182/asheducation-2013.1.82. PMID 24319167
- [Background] Wu Y, Yu J, Zhang L, Luo Q, Xiao JW, Liu XM, Xian Y, Dai BT, Xu YH, Su YC. [Hematopoiesis support of mesenchymal stem cells in children with aplastic anemia]. Zhongguo Dang Dai Er Ke Za Zhi. 2008 Aug;10(4):455-9. Chinese. PMID 18706160
- [Background] Couban S, Simpson DR, Barnett MJ, Bredeson C, Hubesch L, Howson-Jan K, Shore TB, Walker IR, Browett P, Messner HA, Panzarella T, Lipton JH; Canadian Bone Marrow Transplant Group. A randomized multicenter comparison of bone marrow and peripheral blood in recipients of matched sibling allogeneic transplants for myeloid malignancies. Blood. 2002 Sep 1;100(5):1525-31. doi: 10.1182/blood-2002-01-0048. PMID 12176866
- [Background] Watanabe T, Takaue Y, Kawano Y, Koike K, Kikuta A, Imaizumi M, Watanabe A, Eguchi H, Ohta S, Horikoshi Y, Iwai A, Makimoto A, Kuroda Y; Peripheral Blood Stem Cell Transplantation Study Group of Japan. HLA-identical sibling peripheral blood stem cell transplantation in children and adolescents. Biol Blood Marrow Transplant. 2002;8(1):26-31. doi: 10.1053/bbmt.2002.v8.pm11846353.